CLINICAL TRIAL: NCT01866605
Title: A Study of Methods to Reduce Anxiety in Preoperative Elective Surgical Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HREC 2008.074
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2009-02

CONDITIONS: Anxiety
Keywords: anxiety; midazolam; forced-air warming
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): Single un-warmed cotton blanket over body and limbs, and reassurance, during preoperative period in anaesthetic room
  Interventions: Drug: Normal Saline
- 2 (Active Comparator): Single un-warmed cotton blanket over body and limbs, reassurance and intravenous midazolam 30 µg/kg i.v, during preoperative period in anaesthetic room
  Interventions: Drug: Midazolam
- 3 (Active Comparator): Single un-warmed cotton blanket, reassurance and forced-air warming with a Bair Hugger, during preoperative period in anaesthetic room
  Interventions: Device: Bair Hugger

INTERVENTIONS:
Drug: Midazolam — Intravenous midazolam 0.3 mg/kg
  Arms: 2
Drug: Normal Saline — Normal saline injection will be given to groups not receiving midazolam
  Arms: 1
Device: Bair Hugger — Forced air warming
  Arms: 3

SUMMARY:
Patients are often anxious immediately before surgery. The investigators hypothesis is that a warming blanket is as effective as the sedative midazolam in allaying anxiety before surgery.

DETAILED DESCRIPTION:
The investigators are randomising patients aged 18-70 having elective surgery to 1) a cotton blanket and reassurance as required; 2) midazolam, a cotton blanket and reassurance as required; and 3) forced-air warming, a cotton blanket and reassurance as required. The primary endpoint is a visual analog scale of anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years
* male and female
* presenting for elective surgery
* requiring general anaesthesia
* ASA 1-3

Exclusion Criteria:

* Cardiothoracic and intracranial surgery
* Day case surgery
* Pre-existing anxiety disorder
* Patients on psychotropic drugs preoperatively Febrile patients T > 37.5 degrees Celsius Allergy to midazolam Obstructive Sleep Apnoea diagnosed on sleep study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Visual analog scale score for anxiety | During immediate pre-operative phase

SECONDARY OUTCOMES:
Thermal comfort | During immediate pre-operative phase
Recovery from anaesthesia | During immediate post-operative phase
Satisfaction with care | During immediate post-operative phase

CONTACTS AND LOCATIONS:
Overall Officials: Kate Leslie, MD, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Parkville, Victoria, Australia